CLINICAL TRIAL: NCT02237508
Title: An Open-Label, Single-dose, Randomized, Five-Period Cross-over to Compare Pharmacokinetics Profiles of Z7200 and Symbicort Turbohaler, With and Without Charcoal Blockade in Healthy Volunteers.
Brief Title: A Clinical Study to Evaluate Z7200 (Budesonide/Formoterol) Pharmacokinetics Profile in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Z7200J02; 2014-002081-69 (EudraCT Number)
Record Dates: First submitted 2014-09-02; First posted 2014-09-11 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Charcoal; Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- A-B1-B2-C-D (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following 5 treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 days followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B1-C-A-D-B2 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- C-D-B1-B2-A (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- D-B2-C-A-B1 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B2-A-D-B1-C (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- D-C-B2-B1-A (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B2-D-A-C-B1 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- A-B2-B1-D-C (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B1-A-C-B2-D (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- C-B1-D-A-B2 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal

INTERVENTIONS:
Drug: Z7200 without oral activated charcoal — 160 ug budesonide and 4.5 ug formoterol fumarate dihydrate, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler (Treatment A).
  Other Names: budesonide/formoterol
Drug: Symbicort Turbohaler without oral activated charcoal — 320 ug budesonide and 9 ug formoterol fumarate dihydrate, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation (Treatments B1 and B2).
  Other Names: budesonide/formoterol
Drug: Z7200 with oral activated charcoal — 160 ug budesonide and 4.5 ug formoterol fumarate dihydrate, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler with a charcoal blockade (Treatment C).
  Other Names: budesonide/formoterol with coadministration of charcoal
Drug: Symbicort Turbohaler with oral activated charcoal — 320 ug budesonide and 9 ug formoterol fumarate dihydrate, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation from a Symbicort Turbohaler, with charcoal blockade (Treatment D).
  Other Names: budesonide/formoterol with coadministration of charcoal

SUMMARY:
The primary objective was:

- to assess the bioequivalence of a single dose (two inhalations) of the test product compared to the reference product, with and without charcoal blockade.

The secondary objectives were:

* to assess the pharmacokinetic profile of budesonide and formoterol in plasma after a single dose (two inhalations) of the test product and the reference product, with and without charcoal blockade.
* to assess the safety and tolerability of the test product and the reference product, with and without charcoal blockade.

DETAILED DESCRIPTION:
This was a single center, open label, randomized, five-period crossover, single-dose study in healthy volunteers aged 18 to 45 years. A total of 90 volunteers were enrolled, with 9 subjects in each of the 10 treatment sequences.

The study consisted of 5 treatment periods, each lasting approximately 48h, separated by a washout period of a minimum of 5 days. RS01 and/or Symbicort Turbohaler device use training was provided on Day -1 and Day 1 of each treatment period. Subjects were screened for eligibility to participate in the study -28 to -2 days prior to the first treatment period, and were randomized to one of 10 treatment sequencies containing the following 5 treatment arms on Day 1 of the first treatment period:

Treatment A: Z7200 without oral activated charcoal* Treatment B1: Symbicort 1 without oral activated charcoal* Treatment B2: Symbicort 2 without oral activated charcoal* Treatment C: Z7200 with oral activated charcoal** Treatment D: Symbicort with oral activated charcoal**

Subjects were admitted to the clinical unit at 8.00 on the morning of Day -1, and were dosed on the morning of Day 1 following an overnight fast (minimum of 8h). On Day 2, following collection of the 24-h PK blood sample, subjects were discharged.

* Subjects who received treatments A, B1 and B2 rinsed their mouth vigorously with 50 mL water for 3 to 5 sec immediately after the second inhalation.

** A charcoal blockade was used to prevent absorption from oropharyngeal and GI tract, in order to assess the pulmonary deposition of budesonide and formoterol, with periods performed without a charcoal blockade allowing the assessment of the total systemic exposure to the drug.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female 18 to 45 years of age.
* If female, is currently not pregnant/breast feeding/ or attempting to become pregnant has a negative serum pregnancy test, or is of non-childbearing potential or is of child-bearing potential, willing to commit to using a consistent and acceptable method of birth control or is of child-bearing potential and not sexually active
* Body mass index (BMI) of 18.5 to 29.9 kg/m² inclusive and a body weight ≥50 kg.

Main Exclusion Criteria:

* FEV1 value less than 80% of the predicted value and FEV1/FVC ratio <0.7.
* History or current evidence of a clinically significant disease or disorder capable of altering the absorption, metabolism, distribution or elimination of drugs.
* History or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, haematological, neuropsychological, endocrine, gastrointestinal or pulmonary.
* Presence of glaucoma, cataracts, ocular herpes simplex, malignancy, regardless of the clinical significance or current stability of the disease.
* History or presence of silent infections, including positive tests for HIV1, HIV2, Hepatitis B and Hepatitis C.
* Bacterial or viral infection of the upper respiratory tract (including the common cold and flu), sinus, or middle ear within 2 weeks of dosing.
* Lower respiratory tract infection/pneumonia within the past 3 months.
* Presence of any disease or condition or regular concomitant treatment (including vitamins and herbal products) known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Screening haemoglobin value of less than 1g/dL above the ULN (or 10g/L)
* History of recurrent vasovagal collapses.
* History of anaphylactic/anaphylactoid reactions.
* History of seizures including febrile seizures excluding childhood febrile convulsions.
* Unable to demonstrate proper inhalation techniques involved in using the delivery devices at screening.
* Exposure to any investigational drug within 90 days of the Screening Visit.
* Known or suspected hypersensitivity or idiosyncratic reaction to any steroid, any β2 agonist,or to lactose monohydrate, leucine or Tween 80.
* History of allergy to milk protein.
* Use of an inhaled corticosteroid within 30 days or systemic corticosteroid within 60 days of the Screening Visit.
* Use of medications or herbal medicines that are strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers within 30 days prior to Screening Visit
* Any clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study.
* Use of caffeine containing beverages more than 600 mg of caffeine/day.
* Current smokers or ex-smokers who have stopped smoking for less than 10 years.
* Recent or current (suspected) drug abuse or positive result in the drugs abuse test.
* Recent or current alcohol abuse (regular drinking more than 21 units per week for males and more than 14 units per week for females [1 unit = 4 cl spirits or equivalent]).
* Predictable poor compliance, intolerance to charcoal solution, or inability to communicate well with the study centre personnel or inability to participate in all treatment periods.
* The subject is not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions, has participated in a clinical research study within the previous three months or has previously been enrolled in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Evans, MBChB, Principal Investigator — Quotient Clinical Limited
Locations (1):
- Quotient Clinical Ltd, Ruddington, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened for eligibility -28 to -2 days prior to the first treatment period. On Day -1 of the first treatment period, i.d. before randomization, subjects were trained on both the RS01 and Symbicort Turbohaler devices.
Pre-assignment Details: Subjects had to have an adequate inspiratory flow rate and be able to use both inhalers. Subjects who continued to meet all entry criteria on Day -1 of treatment Period 1 and with an inspiratory flow rate of ≥60 L/min and proper device use entered the treatment phase.
Groups:
- A-B1-B2-C-D; B1-C-A-D-B2; C-D-B1-B2-A; D-B2-C-A-B1; B2-A-D-B1-C; D-C-B2-B1-A; B2-D-A-C-B1; A-B2-B1-D-C; B1-A-C-B2-D; C-B1-D-A-B2: Subjects were dosed on Day 1 of each treatment period with one of the following 5 treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B1: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period ≥5 days followed treatment periods 1 to 4.
  Z7200 without activated charcoal: 160 ug budesonide and 4.5 ug formoterol, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler (Treatment A).
  Symbicort Turbohaler without activated charcoal: 320 ug budesonide and 9 ug formoterol, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation (Treatments B1 and B2).
  Z7200 with activated charcoal: 160 ug budesonide and 4.5 ug formoterol, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler with a charcoal blockade (Treatment C).
  Symbicort Turbohaler with activated charcoal: 320 ug budesonide and 9 ug formoterol, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation, with charcoal blockade (Treatment D).
Period: Overall Study
Arm/Group | A-B1-B2-C-D | B1-C-A-D-B2 | C-D-B1-B2-A | D-B2-C-A-B1 | B2-A-D-B1-C | D-C-B2-B1-A | B2-D-A-C-B1 | A-B2-B1-D-C | B1-A-C-B2-D | C-B1-D-A-B2
Started | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
A | 9 | 6 | 8 | 8 | 9 | 8 | 8 | 9 | 9 | 9
B1 | 9 | 9 | 9 | 8 | 9 | 9 | 9 | 9 | 9 | 9
B2 | 9 | 6 | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
C | 9 | 8 | 9 | 8 | 9 | 9 | 9 | 9 | 9 | 9
D | 9 | 6 | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
Completed | 9 | 6 | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 9
Not Completed | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All subjects who received at least one dose (2 inhalations) of investigational medicinal product.
Groups:
- Total: Total of all reporting groups
Arm/Group | A-B1-B2-C-D | B1-C-A-D-B2 | C-D-B1-B2-A | D-B2-C-A-B1 | B2-A-D-B1-C | D-C-B2-B1-A | B2-D-A-C-B1 | A-B2-B1-D-C | B1-A-C-B2-D | C-B1-D-A-B2 | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 90
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (7.9) | 24.7 (6.5) | 27.2 (6.0) | 28.1 (7.4) | 26.3 (7.6) | 29.8 (8.5) | 28.0 (7.6) | 28.3 (5.9) | 27.8 (8.9) | 36.2 (5.0) | 28.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 1 | 2 | 5 | 5 | 3 | 5 | 4 | 37
  Male | 6 | 4 | 5 | 8 | 7 | 4 | 4 | 6 | 4 | 5 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 5
  White | 7 | 9 | 9 | 9 | 8 | 8 | 7 | 9 | 8 | 6 | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 90

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t of Budesonide With and Without Charcoal Blockade
Description: Area under the plasma concentration-time curve from time zero to the last detectable level calculations were performed using the linear trapezoidal rule.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: PK population included subjects who had received both test and reference for at least one dose of each treatment without or with oral charcoal.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Treatment A: Z7200 without charcoal (160 ug budesonide)
- Treatment B: Symbicort 1+2 without charcoal (320 ug budesonide)
- Treatment C: Z7200 with charcoal (160 ug budesonide)
- Treatment D: Symbicort with charcoal (320 ug budesonide)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
pg*h/mL | 1870 (20.2) | 1360 (49.4) | 1810 (22.3) | 1330 (52.3)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — Z7200 was considered bioequivalent to the reference if the following criteria were satisfied: * the 90%CI for the geometric mean AUC0-t ratio was within the interval 80.00% to 125.00% for both budesonide and formoterol, with and without charcoal blockade and * the 90%CI for the geometric mean ratio for Cmax was within the wider bioequivalence acceptance limits of (69.84%, 143.19%) for budesonide and (71.92%, 139.04%) for formoterol, respectively with and without charcoal blockade; p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 138.87, 90% CI 2-sided [129.09 to 149.39]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 136.18, 90% CI 2-sided [126.13 to 147.04]

2. Primary Outcome: AUC0-t of Formoterol With and Without Charcoal Blockade
Description: as for outcome 1
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Treatment A: Z7200 without charcoal (4.5 ug formoterol)
- Treatment B: Symbicort 1+2 without charcoal (9 ug formoterol)
- Treatment C: Z7200 with charcoal (4.5 ug formoterol)
- Treatment D: Symbicort with charcoal (9 ug formoterol)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
pg*h/mL | 47.4 (26.0) | 40.1 (58.6) | 44.7 (26.8) | 34.5 (78.1)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 119.73, 90% CI 2-sided [109.40 to 131.03]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 129.62, 90% CI 2-sided [117.33 to 143.20]

3. Primary Outcome: Cmax of Budesonide With and Without Charcoal Blockade
Description: Maximum plasma level of budesonide with and without charcoal blockade. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
pg/mL | 1040 (67.7) | 482 (63.4) | 1090 (78.9) | 542 (62.4)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 218.13, 90% CI 2-sided [194.02 to 245.24]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 200.66, 90% CI 2-sided [174.30 to 231.01]

4. Primary Outcome: Cmax of Formoterol With and Without Charcoal Blockade
Description: Maximum plasma level of formoterol with and without charcoal blockade. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
pg/mL | 11.9 (38.6) | 9.53 (57.5) | 12.4 (35.5) | 10.6 (58.4)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 126.17, 90% CI 2-sided [115.93 to 137.32]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.004, Mixed Models Analysis; Adjusted geometric means ratio = 117.08, 90% CI 2-sided [107.05 to 128.05]

5. Secondary Outcome: AUC0-30 of Budesonide With and Without Charcoal Blockade.
Description: Area under the plasma concentration-time curve from time zero to 30 minutes calculations were performed using the linear trapezoidal rule.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-30 min (0, 2, 5, 10, 15, 20, and 30 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
pg*h/mL | 324 (36.5) | 174 (62.0) | 342 (38.3) | 193 (63.4)

6. Secondary Outcome: AUC0-30 of Formoterol With and Without Charcoal Blockade.
Description: as for outcome 5
Time Frame: 0-30 min (0, 2, 5, 10, 15, 20, and 30 min)
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
pg*h/mL | 3.85 (33.0) | 3.12 (54.4) | 4.00 (32.1) | 3.35 (58.2)

7. Secondary Outcome: AUC0-∞ of Budesonide With and Without Charcoal Blockade
Description: Area under the plasma concentration-time curve from time zero to infinity calculations were performed using the linear trapezoidal rule.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 163 | 84 | 84
pg*h/mL | 1980 (20.5) | 1450 (48.8) | 1900 (22.4) | 1410 (50.1)

8. Secondary Outcome: AUC0-∞ of Formoterol With and Without Charcoal Blockade
Description: as for outcome 7
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 61 | 126 | 75 | 63
pg*h/mL | 56.0 (28.2) | 49.8 (57.1) | 54.5 (27.7) | 45.2 (61.6)

9. Secondary Outcome: Tmax for Budesonide With and Without Charcoal Blockade
Description: Time at which the maximum plasma level (Cmax) occurred with and without charcoal blockade.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
hours | 0.08 [0.03 to 0.75] | 0.25 [0.03 to 1.50] | 0.08 [0.03 to 0.75] | 0.25 [0.03 to 1.00]

10. Secondary Outcome: Tmax for Formoterol With and Without Charcoal Blockade
Description: as for outcome 9
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 164 | 84 | 84
hours | 0.08 [0.08 to 0.20] | 0.08 [0.04 to 0.25] | 0.08 [0.03 to 0.17] | 0.08 [0.08 to 0.17]

11. Secondary Outcome: t1/2 for Budesonide With and Without Charcoal Blockade
Description: Apparent elimination half-life calculated as 0.693/lambda zeta, with and without charcoal blockade.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 163 | 84 | 84
hours | 2.90 (17.0) | 2.94 (19.8) | 2.79 (17.0) | 2.80 (15.8)

12. Secondary Outcome: t1/2 for Formoterol With and Without Charcoal Blockade
Description: as for outcome 11
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 61 | 126 | 75 | 63
hours | 9.57 (29.3) | 9.33 (35.2) | 10.09 (29.8) | 9.15 (33.6)

13. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 refers to the volume of air that an individual can exhale during a forced breath in 1 second.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
  and Symbicort 2, together. Please note that, within the safety population, 90 subjects received Treatment B. This would mean that theorically 180 participants received Symbicort 1 and Symbicort 2, together.
  But some subjects were excluded from the statistical analysis for various reasons so that the total number included in the statistical anlysis for treatment B is 174.
Time Frame: At 75 min (1.25 hours) post-dose
Population: Safety population: all subjects who received at least one dose (2 inhalations) of investigational medicinal product
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Treatment A: Z7200 without charcoal
- Treatment B: Symbicort 1+2 without charcoal
- Treatment C: Z7200 with charcoal
- Treatment D: Symbicort with charcoal
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 84 | 174 | 87 | 86
liters | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.2)

14. Secondary Outcome: Change From Baseline in the Ratio of Forced Expiratory Volume in 1 Second to Forced Vital Capacity (FEV1/FVC)
Description: FVC = Forced vital capacity. It is the full amount of air that can be exhaled with effort in a complete breath.
  FEV1/FVC = Tiffenau-Pinelli Index. This parameter represents the measurement of the amount of air an individual can forcefully exhale from his/her lungs.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
  Please note that, within the safety population, 90 subjects received Treatment B. This would mean that theorically 180 participants received Symbicort 1 and Symbicort 2, together.
  But 6 subjects were excluded from the statistical analysis for various reasons so that the total number included in the statistical anlysis for treatment B is 174.
Time Frame: At 75 min (1.25 hours) post-dose
Population: Safety population: all subjects who received at least one dose (2 inhalations) of investigational medicinal product.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 84 | 174 | 87 | 86
ratio | 3.7 (3.0) | 3.6 (3.4) | 3.2 (3.1) | 3.8 (3.2)

15. Secondary Outcome: Change From Baseline in Peak Expiratory Flow Rate (PEFR)
Description: PEFR is the highest rate at which gases can be expelled from the lungs via an open mouth. Its measurement is a simple procedure in which an individual takes a full inspiration and blows out as forcibly as possible into an instrument called a peak flow meter, which measures the maximal gas flow in an exhalation in liters per minute.
  Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.Please note that, within the safety population, 90 subjects received Treatment B. This would mean that theorically 180 participants received Symbicort 1 and Symbicort 2, together. But 6 subjects were excluded from the statistical analysis for various reasons so that the total number included in the statistical anlysis for treatment B is 174.
Time Frame: At 75 min (1.25 hours) post-dose
Population: Safety population: all subjects who received at least one dose (2 inhalations) of investigational medicinal product.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 84 | 174 | 87 | 86
L/min | 22.2 (48.9) | 20.5 (38.7) | 24.8 (35.5) | 19.2 (38.9)

ADVERSE EVENTS:
Time Frame: Throughout the study till the end of trial assessment, which was completed on Day 2 of last treatment period (up to 6 weeks).
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/90 | 0/88 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/90 | 0/88 | 0/86
Other Adverse Events (participants affected / at risk) | 16/84 | 20/90 | 6/88 | 15/86
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=84) | Treatment B (N=90) | Treatment C (N=88) | Treatment D (N=86)
Headache (Nervous system disorders) | 5 (5) | 8 (8) | 2 (2) | 7 (7)
Migrane (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations and Caveats not specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No